## **BDF ROYAL MEDICAL SERVICES**



## **Patient Consent for Publication of Materials in BDFRMS**

The following information must be provided for this form to be processed accurately.

File No:

| Author(s): Dr. Mehtash butt, Dr. Jalal. Patients have the right to refuse to sign this consent forum; recare in anyway | fusal to sign this form will not affect their |
|---|---|
| I hereby give my consent for images or other clinical inform BDF Royal Medical Services | nation relating to my case to be used by |
| I understand that my name and initials will not be published and that efforts will be made to conceal m identity, but that anonymity cannot be guaranteed. | |
| I understand that the material may be utilized by BDFRMS may be seen by the general public. I understand that the mapublished by IN House Training. | |
| Name of the Patient | Patient's date of Birth |
| Signature of patient (or signature of the Person giving consent on behalf of the patient) | Date |
| If you are not the patient, what is your relationship to him of a substitute decision maker or legal guardian or should hold | |
| Why is the patient not able to give consent? (e.g.; is the pati | ent a minor, incapacitated, or deceased?) |
| If images of the patient's face or distinctive body markings arbe signed in addition to the first section: | e to be published, the following section should |
| De digned in addition to the mist be circuit | markings to be published and recognize that |

Please complete all required fields (file number, title and author) before returning to: PO. Box 28743, Riffa or by mail: <a href="mailto:training.directorate@bdfmedical.org">training.directorate@bdfmedical.org</a> or fax: 17766822

Date:

Signature of patient (or signature of the persons giving

Consent on behalf of the patient)